CLINICAL TRIAL: NCT02490553
Title: ELISABET : Enquête LIttoral Souffle Air Biologie Environnement
Brief Title: Epidemiological Study on the Relationship Between Respiratory Health and Air Pollution From Industrial Sources
Acronym: ELISABET
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_32/1003; 2010-A00065-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-06-25; First posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Airway Obstruction; Hypertension; Diabetes Mellitus; Dyslipidemias; Pulmonary Disease, Chronic Obstructive
Keywords: air pollution; epidemiological survey; representative sample
MeSH Terms: conditions — Airway Obstruction; Hypertension; Diabetes Mellitus; Dyslipidemias; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * A 2 ml aliquot of heparinized plasma stored at -20 ° C
  * Five 0.5 ml aliquots of EDTA plasma stored at -80 ° C
  * Two 1-ml aliquots of EDTA blood stored at -80 ° C
  * An aliquot of 10 ml and three aliquots of 5 ml of urine stored at -80 ° C
  * Two locks of hair preserved in an envelope at room temperature
  * Six 0.250 ml aliquots of condensate stored at -80 ° C
  * DNA extraction.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dunkirk area: Representative sample of Dunkirk and the surrounding urban area (of ~200 000inhabitants).Dunkirk area is characterize by high emission of industrial air pollutant
  Interventions: Other: heteroevaluation scale by a nurse or doctor
- Lille area: Representative sample of Lille and the surrounding urban area (of ~1 million inhabitants, the fourth urban area in France)
  Interventions: Other: heteroevaluation scale by a nurse or doctor

INTERVENTIONS:
Other: heteroevaluation scale by a nurse or doctor

SUMMARY:
The ELISABET STUDY is across sectional Survey on a representative sample of two urban area conduct on a representative sample. The main objective of the project is to compare the prevalence of the obstructive ventilatory disorders (OVD) in the Urban Community of Dunkirk touched by the industrial pollution in relation to the one recovered in the Urban Community of Lille (CUDL) less industrialized.

DETAILED DESCRIPTION:
Airflow obstruction include Pulmonary Disease, Chronic Obstruction and asthma. Identification of Airflow obstruction is through Functional Tests Lung. In the 1950s, high pollution levels were associated with increased mortality. Despite a reduction of air pollution, it has been established that pollution peaks have short-term effects on acute respiratory episodes. The Urban Community of Dunkirk (CUD) focuses many large pollutant emitters. The long term effects of industrial pollution on TVO are unknown.

The main objective of the project is to compare the prevalence of Airflow obstruction in the Urban Community of Dunkirk affected by industrial pollution compared to that found in the Urban Community of Lille (CUDL) less industrialized. Secondary objectives are: 1) To assess the relationship between air pollution from industrial and biological markers, particularly the plasma concentrations of heavy metals 2) To assess the prevalence of TVO general population in French populations 3) Establish a baseline epidemiological and biological bank.

ELIGIBILITY:
Inclusion Criteria:

* had lived for at least 5 years in the same city or its surrounding urban area (either Lille or Dunkirk) in the northern of France
* Agreed to participate and signed contentment

Exclusion Criteria:

* The detainees
* People under legal protection
* Individuals unable to consent

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants were selected from electoral rolls by random sampling, with stratification for gender, age and centercentre (Lille or Dunkirk). All participants were all recruited between January 2011 and November 2013. Each selected participant received a letter asking him/her to contact the coordinating team and make an appointment for data collection. In the absence of a reply, participants were contacted by telephone. Data was collected at home (occasionally during a consultation in a healthcare establishment). In all cases, a trained, registered nurse administered a detailed questionnaire and performed spirometry testing.
Sampling Method: Probability Sample
Enrollment: 3276 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
airway obstruction | during a the single visit scheduled (less than 3 hours in the morning)
  Forced expiratory volume per second (FEV1) to forced vital capacity (FVC) ratio below 0.7. mesured by standardized spirometry
  Spirometry testing was performed mostly at home using Micro 6000 spirometers (Medisoft; Sorinnes, Belgium), according to the 2005 ATS/ERS guidelines. The spirometers were calibrated weekly. No bronchodilators were administered. For each participant, the spirometry test was repeated (up to seven times) until three acceptable, reproducible flow-volume loops were obtained, following the same guidelines. The greatest reproducible values of FEV1 and FVC were selected for the statistical analysis (regardless of whether these two values came from separate curves or from the same curve). All spirometry data were validated by an experienced, specialist physician.

SECONDARY OUTCOMES:
hypertension | during a the single visit scheduled (less than 3 hours in the morning)
  Hypertension was defined as ongoing antihypertensive treatment, an Systolic blood pressure >=140 mmHg or a Diastolic Blood pressure >=90 mmHg
dyslipidemia | during a the single visit scheduled (less than 3 hours in the morning)
  Dyslipidemia was defined as ongoing cholesterol-lowering treatment or one or more abnormal fasting blood lipid values (total cholesterol 2.4 g/L, LDLcholesterol>=1.6 g/L, HDLcholesterol <0.4 g/L or blood triglycerides >=2 g/L)
diabetes mellitus | during a the single visit scheduled (less than 3 hours in the morning)
  Diabetes mellitus was defined as ongoing antidiabetes treatment (oral medication or insulin) or a fasting blood glucose (FBG) level >=1.26 g/L

CONTACTS AND LOCATIONS:
Overall Officials: Luc Dauchet, PhD MD, Principal Investigator — CHRU LILLE